CLINICAL TRIAL: NCT07064655
Title: A Prospective Observational Cohort Study of Patients Undergoing Non-gastric Conduit Reconstruction After Esophagectomy to Assess Surgical Outcomes
Brief Title: Non-gastric Conduit Reconstruction After Esophagectomy
Status: Not yet recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Seong Yong Park, Associate Professor, MD, Ph.D, Department of Thoracic and Cardiovascular Surgery, Samsung Medical Center
Other Study IDs: SMC 2025-05-092
Record Dates: First submitted 2025-07-05; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Esophagectomy; Esophageal Cancer
Keywords: esophageal cancer; esophagectomy; non-gastric conduit reconstruction
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non-gastric conduit group: Patients who received the reconstruction other than a gastric conduit after esophagectomy

SUMMARY:
This study is to collect and analyze the clinical information of patients who underwent reconstruction using conduits other than the stomach, such as the colon and small intestine, after esophagectomy. Currently, reconstruction after esophagectomy is mainly performed using the stomach, and there is very little information on reconstruction using the colon and small intestine.

Therefore, this study aims to collect information on patients who underwent reconstruction using conduits other than the stomach, analyze the surgical performance, find clinical improvements, and build a foundation for future clinical quality improvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have voluntarily signed an informed consent form and are willing and able to complete all requirements of the study.
* Age 20 years or older.
* Patients who are scheduled for esophagectomy and reconstruction with a conduit other than a gastric conduit is planned.

Exclusion Criteria:

* Patients who do not consent to participate in this study
* The investigator determines that the patient should not participate in the study because the investigator believes that the patient will not be able to comply with the study procedures, requirements, and procedures

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients registered at Samsung Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2030-06-15 (Estimated); Study Completion 2030-12-30 (Estimated)

PRIMARY OUTCOMES:
anastomotic leakage rate | From enrollment to 6 months after esophagectomy
rate of conduit necrosis | From enrollment to 6 months after esophagectomy

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) from this study, because the consent form did not include provisions for data sharing and institutional policy does not permit it.